CLINICAL TRIAL: NCT02039167
Title: WATCH Bleeding Episodes After Left Atrial Appendage Occlusion Versus Usual Care in Patients With Atrial FIBrillatIon and Severe to eNd-stage Chronic Kidney Disease (WatchAFIB in CKD)
Brief Title: Left Atrial Appendage Occlusion vs. Usual Care in Patients With Atrial Fibrillation and Severe Chronic Kidney Disease
Acronym: WatchAFIB
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The recruitment rate was very poor. The study was stopped by amendment on 2015-08-28.
Sponsor: University of Magdeburg (Other)
Responsible Party: Principal Investigator, Prof Dr Ruediger C. Braun-Dullaeus, Prof Dr, University of Magdeburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OVGU-014-Kar
Record Dates: First submitted 2014-01-15; First posted 2014-01-17 (Estimated); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Blood Coagulation Disorders; Atrial Fibrillation; Thrombosis of Left Atrial Appendage; Chronic Kidney Disease Stage 4; Chronic Kidney Disease Stage 5
MeSH Terms: conditions — Blood Coagulation Disorders; Atrial Fibrillation; Renal Insufficiency, Chronic | interventions — Left Atrial Appendage Closure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Left atrial appendage occlusion (Active Comparator): Percutaneous left atrial appendage closure using the WATCHMAN device.
  Interventions: Device: Left atrial appendage occlusion
- OAC with a vitamin K antagonist (No Intervention): Oral anticoagulants (OAC) as Standard of Care (SOC) provided by primary care physician

INTERVENTIONS:
Device: Left atrial appendage occlusion — Percutaneous left atrial appendage closure using the WATCHMAN device.
  Arms: Left atrial appendage occlusion

SUMMARY:
The purpose of this study is to evaluate the superiority of left atrial appendage occlusion in comparison to oral anticoagulation with a vitamin K antagonist (INR 2-3) related to the frequency of occurrence of at least one bleeding classified as moderate or major within 24 months.

DETAILED DESCRIPTION:
Open, randomized, controlled, multicenter clinical investigation. Transesophageal echocardiography (TEE) for all patients within 14 days of the Enrolment Visit. Patients randomized to oral anticoagulation (OAC) will receive standard of care (SOC) vitamin K antagonist treatment throughout the 24 months clinical investigation period, managed by the primary care physician, with the goal of achieving and maintaining an INR of 2-3 (INR monitoring by the primary care physician every two weeks throughout study period).

Patients randomized to the WATCHMAN device will undergo device implantation within 48 hours of the screening TEE and after confirmation of INR ≤ 1.7 in the catheterization laboratory with a subsequent hospitalization for 24-48 hours.

Concomitant treatment with Aspirin/Clopidogrel (managed by the patient's primary care physician) will be initiated on the day prior to device implantation, and will be continued for 6 months after the procedure, at which time Clopidogrel will be discontinued; administration of Aspirin will be continued indefinitely.

Follow-up visits for all patients will take place on Day 45, and at Month 6, Month 12 and Month 24 (End of Study). Routine safety and efficacy assessments at each visit will be the same for all patients regardless of treatment group.

Follow-up- visits at day 45, months 6, 12 and 24. Patients randomized to the WATCHMAN device will have additional TEE imaging performed at the Day 45 and Month 6 visits.

An independent Data Monitoring Committee will monitor safety. A blinded and independent Endpoint Committee will evaluate end-points throughout the entire study period.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal, persistent, or permanent non-valvular atrial fibrillation (AF), documented by electrocardiography performed at screening or within the prior 6 months
* Indication for oral anticoagulation as assessed by CHA2DS2-VASc-Score (≥ 2)
* Severe to end-stage chronic kidney disease (eGFR < 30 ml/min as determined by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula)
* 18 to 80 years, inclusive
* Life expectancy of at least 2 years
* Negative pregnancy test for women
* Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent
* Written informed consent

Exclusion Criteria:

* AF due to a reversible cause or a singular occurrence of AF
* Conditions other than AF that require anticoagulation
* Transient ischemic attack or stroke within previous 3 months
* A need for Aspirin (at a dose of > 162.5 mg/day) or for both Aspirin and Clopidogrel/other antiplatelet drugs (daily administration) other than for clinical investigation
* Contraindications or allergies to vitamin K antagonists, Aspirin or Clopidogrel
* Previous closure (surgical, interventional) of the left atrial appendage (LAA)
* Previous closure of atrial septal defect (ASD) / persistent foramen ovale (PFO)
* Active internal bleeding
* Thrombocytopenia (< 100,000 platelets/mm3)
* History of or planned organ transplantation
* Planned Mitra Clip or transcatheter aortic valve implantation (TAVI) intervention
* Planned cardiac surgery
* History of intracranial, intraocular or retroperitoneal bleeding
* Severe GI-bleeding within the last 3 months
* Hemorrhagic gastro-intestinal diseases (e.g., ulcerative colitis)
* History of or condition associated with increased bleeding risk
* Uncontrolled arterial hypertension
* Heparin-induced thrombocytopenia type II
* Known inherited coagulation disorders
* Severe liver dysfunction (spontaneous INR > 1.5) or liver cirrhosis ≥ CHILD B
* Chronic use of non-steroidal anti-inflammatory drugs (NSAIDs)
* Women who are planning to become pregnant, or who are breastfeeding
* Active infection of any kind

Transesophageal echocardiography (TEE) Exclusion Criteria

* Intracardiac thrombus or dense spontaneous echo contrast as visualized by TEE (with use of sonovue in suspicious cases)
* Significant mitral valve stenosis
* Any congenital heart disease, including atrial septal defect
* Pericardial effusion during ECHO assessment of > 2 mm
* Cardiac tumor

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-01; Primary Completion 2017-03-21 (Actual); Study Completion 2017-04-12 (Actual)

PRIMARY OUTCOMES:
Frequency of occurrence of moderate and major bleedings (Type 2 to Type 5 according to the Bleeding Academic Research Consortium (BARC) definitions) | 24 months

SECONDARY OUTCOMES:
Frequency of at least one occurrence of a combined endpoint of moderate or major bleeding and/or severe cardiovascular adverse events (stroke, cardiac infarction, thrombosis, death) | 24 months

OTHER OUTCOMES:
Time to occurrence of first moderate and major bleeding as well as to occurrence of stroke (ischemic or hemorrhagic) according to the modified Rankin scale | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Rüdiger C Braun-Dullaeus, Prof, Principal Investigator — Otto-von-Guericke University Magdeburg Faculty of Medicine
Locations (4):
- Germany (4):
  - Otto-von-Guericke University Magdeburg, Faculty of Medicine, Magdeburg, Saxony-Anhalt
  - Zentralklinik Bad Berka - Klinik für Kardiologie, Bad Berka
  - CCB im Markus Krankenhaus Frankfurt, Frankfurt
  - Medizinische Hochschule Hannover Zentrum Innere Medizin, Abt. Kardiologie und Angiologie, Hanover